CLINICAL TRIAL: NCT02944045
Title: Intérêt de la corticothérapie Dans la Pneumocystose Grave du Patient immunodéprimé Non VIH. Essai Prospectif Multicentrique Randomisé Contrôlé : PIC
Brief Title: Effect of Steroids During Pneumocystis Infection Among Non HIV Immunocompromised Patients
Acronym: PIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P150961; 2016-002275-10 (EudraCT Number)
Record Dates: First submitted 2016-10-17; First posted 2016-10-25 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Pneumocystis; Steroids; Immunocompromised Patient; Hematologic Neoplasms; Immunosuppressive Agents; Neoplasms
MeSH Terms: conditions — Pneumonia, Pneumocystis; Hematologic Neoplasms; Neoplasms | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline serum, same volume as in the Experimental arm.
  Interventions: Drug: Placebo
- Steroids (Experimental): Methylprednisolone intra veinous
  * Day 1 to 5 : 30mg twice per day
  * Day 6 to 10 : 30mg per day
  * Day 11 to 21 : 20mg per day
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone intra veinous
  * Day 1 to 5 : 30mg twice per day
  * Day 6 to 10 : 30mg per day
  * Day 11 to 21 : 20mg per day
  Arms: Steroids
Drug: Placebo — saline serum
  Arms: Placebo

SUMMARY:
Pneumocystis jiroveci pneumonia (PcP) increased in non HIV immunocompromised patients. Mortality remains high for those patients with comorbidities (50% for patients with the most severe Pneumocystis pneumonia). Physiopathology, characteristics and outcome of PcP in non-HIV patients remains different from those in HIV patients. Steroids in HIV patients with PcP has been associated with decreased mortality but in non-HIV patients, adjunctive steroids remains controversy. Some retrospective studies in that field did not find any beneficial effects of steroids ((1mg/kg/jour d'Equivalent Prednisone (EP)). However, all the studies were retrospective, non randomised studies including various underlying disease and severity of PcP was variable. Moreover, dosage and delay of steroids were variable leading difficult to interpret all the results.

The investigators want to demonstrate the beneficial effect of steroid during PcP in non-HiV immunocompromised patients with a double blinded randomised clinical trials comparing adjunctive steroids to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe PcP : 1 / interstitial acute pneumonia with possible or typical criteria for PcP and positive specimen for Pneumocystis jirovecii (excluding PCR) ; or interstitial acute pneumonia with typical criteria for PcP and positive PCR in respiratory specimen. 2/ Arterial pression of Oxygen (PaO2) < 60 mmHg on room air need of 3 L/min oxygen for saturation >92% or tachypnea>30min need of mechanical ventilation for acute respiratory failure.
* Treatment for PcP started for less than 7 days.
* Non-HIV immunosuppression : malignant hematological disease, solid tumor cured for less than 5 years, allogenic stem cell transplant, Steroids (>0.3mg/kg equivalent prednisone for more than 3 weeks or > 20mg/days for more than one months) or other immunosuppressive treatment for more than one months or solid organ transplantation.
* Signed inform consent by patient or relatives
* Health insurance

Exclusion Criteria:

* HIV Serology HIV 1 or 2 positive
* Need of steroid ≥1mg/kg/j equivalent prednisone for another pathology (acute Graft versus Host disease (GVH= for example)
* Contra-indication for steroids
* Pregnancy of breath-feeding
* Denied to participate
* No health insurance
* tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | Day 28
  28 days mortality after the randomisation

SECONDARY OUTCOMES:
Mortality | Day 90
  90 days mortality after the randomisation
Hospital mortality | Day 120
  Mortality at hospital discharge
ICU mortality | Day 90
  For patients admitted to ICU at ICU discharge
Acute respiratory failure | Day 28
  Acute respiratory failure during treatment defined by one of those criteria within 28 days :
  * Increased need of oxygen (more than 9 l/min of high flow nasal oxygen with Inspired Fraction of Oxygen (fiO2) >50%)
  * Admission to ICU after randomisation
  * Need of mechanical ventilation (invasive or non invasive) or high flow nasal oxygen
Duration of mechanical ventilation | Day 28
  Duration of mechanical ventilation invasive and/or non invasive
Occurrence of septic shock | Day 28
  septic shock is defined as need for vasopressor
acute kidney injury | Day 28
  KDIGO score >=1
Hospital acquired infectious disease | Day 28
  Global incidence incidence of infections. Incidence of pulmonary or extra-pulmonary infections.
  Incidence of bacterial, viral and fungal infections. Diagnosis of infectious disease will be defined by the need of treatment.
Hospital length of stay | Day 120
  Hospital length of stay at hospital discharge
ICU length of stay | Day 90
  ICU length of stay at ICU discharge
Duration of Insulin treatment | Day 28
  Insulin treatment is defined :
  * patient without insulin treatment before study : start of insulin therapy
  * patient treated with insulin before study : increased dose (>30%) of insulin

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Lemiale, MD, Principal Investigator — APHP; Elie Azoulay, MD PHD, Study Director — APHP
Locations (1):
- Medical ICU, Paris, France

REFERENCES:
- [Derived] Lemiale V, Resche-Rigon M, Zerbib Y, Mokart D, De Prost N, Wallet F, Perez P, Kouatchet A, Argaud L, Decavele M, Pene F, Seguin A, Megarbane B, Calvet L, Picard M, Rigault G, Mariotte E, Bouadma L, Theodose I, Tamion F, Klouche K, Colin G, Nyunga M, Moreau AS, Azoulay E. Adjunctive corticosteroids in non-AIDS patients with severe Pneumocystis jirovecii pneumonia (PIC): a multicentre, double-blind, randomised controlled trial. Lancet Respir Med. 2025 Sep;13(9):800-808. doi: 10.1016/S2213-2600(25)00125-0. Epub 2025 Jul 10. PMID 40652952